CLINICAL TRIAL: NCT01446185
Title: Treatment Decision Impact of OncotypeDX™ in HR+, N- Breast Cancer Patients
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genomic Health®, Inc. (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A00577-32; 2010-A00577-32 (Other: AFSSAPS identification number)
Record Dates: First submitted 2010-09-01; First posted 2011-10-05 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: HR+, N- or pN1(mi), Her2- breast cancer adjuvant population; Early Breast cancer; Gene Expression; Node-Negative; treatment options; Hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- a HR+, N- or pN1(mi), Her2- breast cancer adjuvant population (Other)
  Interventions: Device: Oncotype DX breast cancer test

INTERVENTIONS:
Device: Oncotype DX breast cancer test — The Oncotype DX breast cancer test measures the expression of 21 genes of an individual tumor to generate an Recurrence Score result that quantifies the magnitude of chemotherapy benefit and the likelihood of recurrence for early-stage breast cancer patients.
  Other Names: Oncotype DX™

SUMMARY:
Primary objective:

Determine the impact of the Oncotype DX Recurrence Score (RS) on the treatment recommendation made (administration of chemotherapy or not, in addition to hormonotherapy) in a HR+, N- or pN1(mi), Her2- breast cancer adjuvant population.

The impact of Oncotype DX on treatment recommendations can be either a decrease in treatment intensity defined as a change in treatment recommendation from chemotherapy plus hormonal therapy to hormonal therapy alone or an increase in treatment intensity defined as a movement from hormonal therapy alone to the addition of chemotherapy to hormonal therapy.

Patients with HR+, N- breast cancer currently represent around 70% of newly diagnosed breast cancers. These are usually good prognosis tumors. However, on the basis of classical clinical and pathological prognostic parameters and markers, the international consensus guidelines recommend treatment with hormone- and chemotherapy in 85-95% of the cases. Considering the natural disease history, such as documented by the EBCTCG meta-analysis, more than 50% of these patients are overtreated, which leads to unnecessary side effects and costs to the health system and to the society.

Oncotype DX appears to be well adapted to therapeutic de-escalation as it targets HR+, N- patients and is performed on fixed paraffin embedded tissue (FPET). It is therefore best adapted to daily clinical practice as it does not necessitate any specific surgical procedure or tissue freezing.

The prognostic and predictive value of Oncotype DX in ER+, N- patients has been validated on three large adjuvant randomized trials (NASBP B-14, NSABP B-20, and the ATAC study). The test has been commercially available in the USA since 2004, and is being used for more than 50% of the HR+ N- patients in this country.

While Oncotype DX has been validated in the USA, it needs to be independently evaluated in France, in the context of the local treatment guidelines and habits, to provide data that are meaningful to the French health system and to the French medical community.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old.
2. Pre- or post- menopausal women with breast adenocarcinoma, confirmed by a pathologist and who underwent surgery, with a maximum of 4 weeks between surgery and the 2nd therapeutic decision with Oncotype DX.
3. HR positive (at least ER+) breast cancer patients (defined by a threshold of 10% of the cells IHC + without N- or pN1(mi), Her2 - (IHC0, 1, 2+ or FISH -)
4. Patients must be eligible to receive adjuvant chemotherapy as defined by a good Karnofsky index, no hematological, cardiological or hepatic contraindications nor any impeding comorbidity.
5. Patients must have given a written informed consent.

Exclusion Criteria:

1. T3 or T4, HR-, N+ (except pN1 (mi) (sn), Her2+ (IHC 3+ or Fish+) patients.
2. Metastatic patients.
3. Patients who cannot give an informed consent.
4. Patients who cannot receive chemotherapy.
5. Patient who participated in another clinical trial and is still in the exclusion period of any other trial.
6. Mentally disabled patient who has no legal responsibility for herself.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
impact of the Oncotype DX Recurrence Score on the treatment recommendation made | Day 15
  The impact of Oncotype DX on treatment recommendations can be either a decrease in treatment intensity defined as a change in treatment recommendation from chemotherapy plus hormonal therapy to hormonal therapy alone or an increase in treatment intensity defined as a movement from hormonal therapy alone to the addition of chemotherapy to hormonal therapy.

SECONDARY OUTCOMES:
Level of confidence of the physicians relating to their treatment recommendation before and after Oncotype DX RS results | Day 15
  The change in physicians' level of confidence in the treatment recommendation will be measured by the change from baseline to follow-up responses.
Physicians' perceptions regarding the utility of the Oncotype DX. | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Joseph GLIGOROV, Principal Investigator — Hôpital TENON
Locations (6):
- France (6):
  - CHRU Besançon, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Centre d'Oncologie Médicale de Gentilly, Nancy
  - Hôpital TENON, Paris